CLINICAL TRIAL: NCT05899101
Title: IMPACT: A Prospective Cohort Study of the Impact of Opioid and Cannabis Exposure on Fetal Growth
Brief Title: The Impact of Opioid and Cannabis Exposure on Fetal Growth
Acronym: IMPACT
Status: Terminated | Type: Observational
Why Stopped: Due to challenges with participant recruitment the propsective study was terminated.
Sponsor: Dr. Laura Gaudet (Other)
Collaborators: University of Ottawa (Other)
Responsible Party: Sponsor-Investigator, Dr. Laura Gaudet, Associate Professor, Queen's University
Organization: Queen's University (Other)
Other Study IDs: CTO 3968
Record Dates: First submitted 2023-05-19; First posted 2023-06-12 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy Related; Substance Use; Fetal Growth Retardation; Placenta Diseases
Keywords: opioid; cannabis; nicotine; opioid agonist therapy
MeSH Terms: conditions — Substance-Related Disorders; Fetal Growth Retardation; Placenta Diseases; Marijuana Abuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Placenta (fresh-frozen), Placenta (FFPE), Cord Tissue (FFPE), Membrane (FFPE), Cord Blood Serum, Cord Blood Plasma, Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (7):
- 1 - Opioid Only: Illicit and/or sustained prescription opioids only (no cannabis use)
- 2 - OAT Only: Opioid agonist therapy (OAT) only (no cannabis use)
- 3 - Opioid and Cannabis: Illicit and/or sustained prescription opioids with concurrent cannabis use
- 4 - OAT and Cannabis: Opioid agonist therapy (OAT) with concurrent cannabis use
- 5 - Nicotine Only: Nicotine users without opioid exposure
- 6 - Cannabis Only: Cannabis-users without opioid exposure
- 7 - Unexposed: Non-substance exposed healthy pregnancies

SUMMARY:
Individually, both opioid and cannabis exposure during pregnancy are associated with changes in fetal growth. The extent to which opioid and cannabis exposure affect fetal growth is unknown. The Investigators hypothesize that the combination of both substances will impact placental function and subsequent fetal growth more severely than either substance alone. The primary objective is to determine the extent to which fetal growth profiles in opioid-exposed pregnancies are influenced by cannabis exposure. This prospective cohort study will consist of opioid-exposed pregnancies and pregnancies without opioid exposure recruited from 5 obstetrical clinics from across Ontario. A total of 546 participants will be recruited.

DETAILED DESCRIPTION:
As cannabis exposure is prevalent in opioid-exposed pregnancies (36-75%), it is vital to understand the potential additive effect of these two concurrent exposures on the development and health of the feto-placental unit. This information would allow for informed decision making about cannabis use and can serve as an important starting point in the design of effective harm reduction strategies in this patient population. From our professional experience, the majority of opioid-using pregnant individuals are motivated to make lifestyle modifications. Eliminating cannabis may be a realistic change these individuals can make to improve outcomes for their infants.

Individually, both opioid and cannabis exposure during pregnancy are associated with altered fetal growth. The extent to which opioid and cannabis exposure affect fetal growth trajectories is unknown. The Investigators postulate that the combination of both substances will impact placental function and subsequent fetal growth more severely than either substance alone. Delineating this relationship may allow for the development of evidence-based harm reduction strategies focused on eliminating cannabis use in opioid-exposed pregnancies to improve fetal growth.

The overarching hypothesis of this research is that opioid exposure compromises placental growth and function, with significant impacts on vascular development, nutrient transport and metabolic signaling, ultimately impacting fetal growth trajectories. The Investigators further propose that the additive effects of cannabis use, extremely common in these pregnancies, may exacerbate this placental dysfunction.

Thus, the primary objective of this study is to determine the extent to which fetal growth profiles in opioid-exposed pregnancies are influenced by cannabis exposure.

The study population will consist of opioid-exposed pregnancies recruited from 5 obstetrical clinics from across Ontario. A total of 546 participants will be recruited.

ELIGIBILITY:
Inclusion Criteria:

1. Participant who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
2. Participant has given written consent after study has been explained according to local regulatory requirements and before any study specific procedures.
3. Age ≥16 years at the time of consent.
4. Singleton pregnancy.
5. Live fetus (documented positive fetal heart beat prior to recruitment)
6. ≥18 0/7 weeks of gestation and documented anatomy ultrasound at the time of consent.
7. No known significant fetal genetic abnormalities (based on genetic testing, if performed).
8. No significant congenital malformations (such as abnormal fetal morphology, abnormal amniotic fluid levels, significant abnormalities in placenta or umbilical cord), as assessed by fetal anomaly ultrasound scan (also known as a level 2 ultrasound or fetal morphology assessment) conducted at or beyond 18 0/7 weeks of gestation.
9. Willing to provide cord blood.
10. Willing to provide placenta.
11. Willing to provide urine sample for drug testing.
12. Plan to reside in the study area at least until delivery.

Exclusion Criteria:

1. Sustained use of substances other than opioids and cannabis, including methamphetamines, benzodiazepines, alcohol, and cocaine. This is defined as any use after the patient is aware that they are pregnant OR as per the discretion of the investigator.
2. Acute or chronic clinically significant abnormality or poorly controlled pre-existent co-morbidities or any other clinical conditions, as determined by physical examination or standard of care laboratory tests, that, in the opinion of the investigator, might confound study results.
3. Known abnormal placentation including accrete, increta and percreta.
4. Any conditions that, in the Investigator's judgement, may interfere with participant's ability to comply with study procedures or receipt of prenatal care, such as behavioural or cognitive impairment or neuropsychiatric illness.
5. Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product.
6. COVID-19 infection being diagnosed within 14 days of consent - recruitment may be delayed until required isolation period is over.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from participating antenatal clinics at five sites across Ontario. Individuals with sustained opioid exposure during pregnancy will be eligible for inclusion into the study. Most individuals who use opioids/OATs in pregnancy smoke cigarettes (>90%). Thus, opioid unexposed groups will also be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Birthweight | At delivery
  The primary outcome of interest is difference in birthweight (grams) between the exposure groups.

SECONDARY OUTCOMES:
Infant length | At delivery
  Infant length at birth (cm) will be compared between the groups.
Incidence of Neonatal Morbidity | From recruitment until 6 weeks postpartum
  The incidence of neonatal morbidity will be compared between the groups. Severe neonatal morbidity (SNM) will be defined as the presence of at least one of the following elements: Apgar score < 4 at 5 min or severe respiratory distress requiring respiratory support, severe neonatal acidosis (cord artery pH < 7.0 or base excess <-12 mmol/L), admission to the neonatal intensive care unit (NICU), cystic periventricular leukomalacia (cPVL), intraventricular haemorrhage (IVH grades III and IV), surgical necrotizing enterocolitis (NEC requiring surgical treatment or peritoneal drainage) or retinopathy of prematurity (ROP≥stage 3).
Length of Stay at Delivery | From admission for delivery until discharge from hospital after delivery
  Length of hospital stay in hours for delivery between the groups. This will be measured from the date of admission to delivery till the date of discharge from the hospital after delivery.
Length of Antepartum Hospital Stay | From admission to discharge for each hospital stay that does not include delivery
  Length of antepartum hospital admissions in hours between the groups. This will be measured from the date of admission to the date of discharge for any maternal hospital admissions before the admission for delivery.
Readmission rates | From discharge from hospital at delivery till 6 weeks postpartum
  Readmission rates between the groups
Placental Weight | At delivery
  Placental weight (grams) between the groups.
Placental gene expression profiles | At delivery
  Placental gene expression profiles related to vascular development, nutrient transport and metabolic signaling between the groups. These will be assessed using RNA sequencing and spatial transcriptomics.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Gaudet, MD, Principal Investigator — Queen's University
Locations (5):
- Canada (5):
  - Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
The objectives of the IMPACT Biobank are to provide a basis for future research on pregnancy and newborn health. The IMPACT consent for Future Research on Stored Biological Samples obtained from Participants is broad enough to support a range of research on fetal growth, pregnancy and the health of mothers and their children. Biobanking is an optional part of the IMPACT study. Participants may decide not to participate in the optional biobanking research and still participate in the main study.
  The IMPACT Biobank is managed in accordance with the principles set forth in:
  * The Canadian Charter of Rights and Freedoms
  * The World Medical Association Declaration of Helsinki: Ethical Principles for Medical Research Involving Human Subjects
  * The Universal Declaration on Bioethics and Human Rights
  * The Tri-Council Policy Statement: Ethical Conduct for Research Involving Humans
  * The Canadian Institutes of Health Research Best Practices for Protecting Privacy in Health Research
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Up to 25 Years
Access Criteria: The IMPACT Biobank Management Committee (IBMC) makes its decisions, including decisions relating to the future direction of the IMPACT Biobank, on the basis of these standards, objectives and the best available scientific evidence. Only research studies that entail, at most, a minimal risk to Participants will be granted access to the IMPACT Biobank.
  The criteria for granting access include:
  * feasibility;
  * scientific value;
  * minimal risk;
  * availability of Material;
  * contribution to the IMPACT Research Study;
  * public health importance to Canadians.
  The IMPACT Biobank is managed on a not-for-profit basis. The IBMC sets access fees with a view to covering the costs of operating the IMPACT Biobank. To help preserve the integrity and volume of the specimens for future users, part of the access fees will pay for the micro-aliquoting of specimens.
URL: https://www.impactresearchstudy.ca/future-research

REFERENCES:
- See also: Study Website — https://www.impactresearchstudy.ca/